Official Title: A Virtual Navigation Intervention to Reduce Behavioral Health Admissions From Rural Emergency Departments (VIBRANT)

NCT04148521

IRB-Approved Date of document: 10/2/22

### Atrium Health Patient Information Sheet

# Study Title: A Virtual Navigation Intervention to Reduce Behavioral Health Admissions from Rural Emergency Departments (VIBRANT)

## Principal Investigator (Study Doctor): Edwin Wayne Sparks, Jr., MD (704) 631-1654

Dr. Edwin Wayne Sparks is inviting you to participate in a research study examining the benefits of virtual navigation. We want to offer you access to a program available through Atrium Health. The name of the program is Behavioral Health Virtual Patient Navigation. We have licensed clinicians that will provide support and help you navigate a successful transition out of the ED.

Before you decide whether or not to participate in this program, it is important for you to understand why the research is being done and what it will involve. Please take the time to read the following information carefully:

1. What is the purpose of this program? The purpose of this program is to help you successfully transition out of the emergency department. We can help you schedule follow-up appointments, find new providers and connect you with community resources as appropriate. We provide follow-up calls for 45 days and you will have our direct number to contact us as needed.

#### 2. Why have I been invited to participate in this program?

You are eligible to participate in this program because you had a consult with a psychiatrist.

3. What if I don't want to take part in this program, or if I want to withdraw later?

Participation in this program is voluntary. It is completely up to you whether or not you wish to participate. If you decide not to participate, it will not affect your relationship with Atrium Health or any of your doctors. If you wish to withdraw from the program once it has started, you can do so at any time.

#### 4. What does this program involve?

If you agree to participate in this program, we provide follow-up calls for 45 days and you will have our direct number to contact us as needed. Your medical record will be used to determine if the program was beneficial.

### 5. How is this program being paid for?

The program is being sponsored by the Duke Foundation. None of the doctors asking you to participate in this study have received or will receive money or other benefits for personal use. However, the sponsor will give money or other benefits to a research fund, foundation, educational institution, or other organization with which the doctor or study staff is associated.

#### 6. Are there risks to me in taking part in this program?

There are no foreseen physical or psychological risks associated with this study.



#### 7. Will I benefit from the program?

Taking part in this research study may or may not benefit you personally, but researchers may learn new things that will help improve future treatment of patients with a psychiatric consult in the emergency department.

#### 8. Will taking part in this program cost me anything, and will I be paid?

There is no financial cost to you to participate in this study. You will not be paid for participating in this study.

#### 9. What happens with the results?

The records of this study will be confidential. In any report we publish, we will not include any information that will make it possible to identify you. Any references to your identity will be removed prior to reports and/or publications.

#### 10. Who should I contact if I have questions or concerns about the program?

Please contact the program coordinator, Amy Barrett at Amy.Barrett@AtriumHealth.org or by phone at

Thank you for taking the time to consider this program.

This information sheet is for you to keep.